CLINICAL TRIAL: NCT06167239
Title: Effect of Ventilator Trigger Sensitivity Adjustment Versus Threshold Inspiratory Muscle Training on Arterial Blood Gases in Mechanically Ventilated Patients, a Randomized Clinical Trail
Brief Title: Ventilator Trigger Sensitivity Adjustment Versus Threshold Inspiratory Muscle Training on Arterial Blood Gases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, El-Sayed Essam, Lecturer at Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004784
Record Dates: First submitted 2023-11-12; First posted 2023-12-12 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Guillain-Barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Threshold inspiratory muscle trainer (Experimental): Training of the inspiratory muscles by threshold inspiratory muscle trainer.
  Interventions: Other: Threshold inspiratory muscle trainer or ventilator pressure setting inspiratory muscle training techniques
- Ventilator pressure setting inspiratory muscle training (Experimental): Training of the inspiratory muscles by ventilator pressure setting.
  Interventions: Other: Threshold inspiratory muscle trainer or ventilator pressure setting inspiratory muscle training techniques
- Traditional treatment (No Intervention): Only prescribed medical treatment programme

INTERVENTIONS:
Other: Threshold inspiratory muscle trainer or ventilator pressure setting inspiratory muscle training techniques — New techniques to train inspiratory muscles in mechanically ventilated patients
  Arms: Threshold inspiratory muscle trainer; Ventilator pressure setting inspiratory muscle training

SUMMARY:
The aim of the current study is to compare the effect of ventilator trigger sensitivity adjustment versus threshold inspiratory muscle training on arterial blood gases in mechanically ventilated patients.

DETAILED DESCRIPTION:
Failed extubations are not uncommon in most ICUs, the failure rate ranging from 2 to 20%. Since failed extubation is associated with greater hospital morbidity and mortality and longer length of stay, it is imperative to identify screening techniques that minimize the number of failed extubations.

Many studies have been done on the effect of IMT by threshold IMT and adjustment of mechanical ventilator trigger separately, thereby, it is rational to compare between two methods of training to know which is more effective to help in weaning process through its effect on ABGs.

ELIGIBILITY:
Inclusion Criteria:

1. Difficult to wean Guillain barre patients who have been on MV for at least 48 hours. Difficult to wean subjects have been defined as those who fail the first spontaneous breathing trial (SBT)and may require up to 3 SBTs or up to 7 d from the first attempt to achieve successful weaning (B´eduneau G. et al.,2017) and (Annia F. et al.,2019).
2. Age: >18 years.
3. Both sexes will be included.
4. Ventilator mode: Pressure support mode with FiO2≤ 0.5, positive end expiratory pressure (PEEP) will be<8-10cm/H2Oand respiratory rate < 25.
5. Conscious oriented patient with Glasgow coma score ≥13.
6. Alertness will be titrated to a Riker Sedation Agitation Score of 4.
7. PH>7.25, arterial oxygen saturation >90%.
8. Cardiovascular stability.
9. Maximal inspiratory pressure from 15 to 30 cm H2O and able to trigger spontaneous breaths on ventilator.

Exclusion Criteria:

1. Persistent hemodynamic instability as life threatening arrhythmias, acute heart failure.
2. Severe breathlessness, when spontaneously breathing.
3. Any progressive neuromuscular disease that would interfere with responding to inspiratory muscle training (non-stationary course).
4. Spinal cord injury.
5. Skeletal pathology (scoliosis, flail chest, spinal instrumentation) that would seriously impair the movement of the chest wall and ribs.
6. Patients on heavy sedation and respiratory muscle paralysis.
7. High peak airway pressure (barotraumas).
8. BMI ≥ 40.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
PH | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  To measure PH
PaO2 | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  To measure partial pressure of oxygen
PaCO2 | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  To measure partial pressure of carbon dioxide
HCO3 | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  To measure bicarbonate

SECONDARY OUTCOMES:
Rapid shallow breathing index | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  To measure respiratory endurance
The Horowitz index | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  To measure PaO2 /FiO2 ratio
Glasgow coma scale | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  To measure level of consciousness
Riker Sedation-Agitation Scale | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  Arousal/sedation assessment
Respiratory rate | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  Number of breath cycles per minute
Minute ventilation | Pre intervention and immediate post intervention, through study completion, an average of two weeks
  The amount of air that enters the lungs per minute.
Weaning success rate | post intervention at the end of the study, an average of two weeks
  Number of patients weaning from MV

CONTACTS AND LOCATIONS:
Overall Officials: Elmasry, Study Director — Cairo University
Locations (1):
- Kasr Al Ainy School of Medicine, Cairo, Egypt